CLINICAL TRIAL: NCT00120276
Title: Randomized Evaluation of a Surgical Treatment for Off-Pump Repair of the Mitral Valve (RESTOR-MV)
Brief Title: RESTOR-MV: Randomized Evaluation of a Surgical Treatment for Off-Pump Repair of the Mitral Valve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myocor (Industry)
Responsible Party: Myocor, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020202
Record Dates: First submitted 2005-07-07; First posted 2005-07-15 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Mitral Valve Regurgitation; Left Ventricular Dysfunction; Heart Failure
Keywords: Functional Mitral Regurgitation (FMR); Ischemic Mitral Regurgitation; Less invasive repair; Surgical MV repair; Mitral Valve Repair; Heart Failure; Left Ventricular Dysfunction
MeSH Terms: conditions — Mitral Valve Insufficiency; Ventricular Dysfunction, Left; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Less invasive mitral valve repair

SUMMARY:
The purpose of this prospective, randomized, multi-center, pivotal trial is to compare the safety and effectiveness of the off-pump, closed heart Coapsys System (Myocor, Inc.) to open surgical repair of the mitral valve using an annuloplasty ring or band in patients with moderate to severe functional mitral regurgitation.

DETAILED DESCRIPTION:
Patient clinical evaluations will consist of 3-month, 6-month, and 12-month follow up of the primary endpoints. Additional follow up of 18-month, 24-month, and annually thereafter will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2, 3, or 4 functional mitral valve regurgitation per 2D echocardiography
* Patient undergoing concomitant coronary artery bypass graft surgery, either on-pump or off-pump
* Left ventricular ejection fraction greater than or equal to 25%
* Age between 18 and 80 years, inclusive
* Patient is willing and available to return for study follow up
* Ability of the patient or legal representative to understand and provide signed consent for participating in the study.

Exclusion Criteria:

* Structural abnormality of the mitral valve (e.g. calcification or thickening of the valve leaflets, ruptured papillary muscle, ruptured chordae tendinae, mitral valve prolapse, mitral stenosis, etc.)
* Asymptomatic Grade 2 MR (those with NYHA Class < II AND LVEF > 40%)
* Organic valve disease resulting in insufficiency or stenosis of the aortic, pulmonary or tricuspid valve requiring surgical intervention
* Transmural myocardial infarction within 30 day period prior to surgical placement of Coapsys
* NYHA class IV
* Left ventricular end diastolic diameter > 7.0 cm
* Cardiac surgery on an emergency or salvage basis
* Left atrial or left ventricular thrombus
* Left ventricular aneurysm
* Previous mitral valve surgery or other previous cardiac surgery that would preclude proper placement of the Coapsys
* Chronic renal failure requiring dialysis
* Open chest surgery contraindication (e.g., acute respiratory distress, endocarditis, myocarditis, pericarditis)
* Active infection
* Life expectancy of less than 24 months due to conditions other than their cardiac status
* Participation in another investigational drug or device protocol
* Abnormal coronary or cardiac anatomy such that the device could not be placed without interfering with those anatomical structures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Primary effectiveness endpoint to compare the mean change in MR grade in the Coapsys group to the open-heart annuloplasty group from baseline to 12 months. | 12- months
The primary safety endpoint is to compare the rate of primary adverse events (PAE's) through 12 months in the Coapsys group to the PAE rate in the open-heart annuloplasty group. | 12- months

SECONDARY OUTCOMES:
Compare heart failure symptoms, left ventricular geometry, change in MR and TR, adverse events, and hospitalization time and costs of Coapsys group to control group | 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Prairie Research and Education Group, Springfield, Illinois
  - St. Joseph's Mercy Hospital, Ann Arbor, Michigan
  - Covenant Healthcare, Saginaw, Michigan
  - Nebraska Heart Institute, Lincoln, Nebraska
  - New York University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - VA Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Grossi EA, Woo YJ, Patel N, Goldberg JD, Schwartz CF, Subramanian VA, Genco C, Goldman SM, Zenati MA, Wolfe JA, Mishra YK, Trehan N. Outcomes of coronary artery bypass grafting and reduction annuloplasty for functional ischemic mitral regurgitation: a prospective multicenter study (Randomized Evaluation of a Surgical Treatment for Off-Pump Repair of the Mitral Valve). J Thorac Cardiovasc Surg. 2011 Jan;141(1):91-7. doi: 10.1016/j.jtcvs.2010.08.057. PMID 21168015
- [Derived] Grossi EA, Patel N, Woo YJ, Goldberg JD, Schwartz CF, Subramanian V, Feldman T, Bourge R, Baumgartner N, Genco C, Goldman S, Zenati M, Wolfe JA, Mishra YK, Trehan N, Mittal S, Shang S, Mortier TJ, Schweich CJ Jr; RESTOR-MV Study Group. Outcomes of the RESTOR-MV Trial (Randomized Evaluation of a Surgical Treatment for Off-Pump Repair of the Mitral Valve). J Am Coll Cardiol. 2010 Dec 7;56(24):1984-93. doi: 10.1016/j.jacc.2010.06.051. PMID 21126639